CLINICAL TRIAL: NCT06361524
Title: Longitudinal Gut Microbiome and Host Multi-omic Profiling in Patients With Chronic Heart Failure
Brief Title: Gut Microbiome Profiling in Patients With Chronic Heart Failure
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Petra Mamic, Instructor, Stanford University
Other Study IDs: 44967; 5F32HL143916 (NIH); 856341 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-04-05; First posted 2024-04-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Nonischemic Cardiomyopathy
Keywords: Gut microbiome; Gut microbiota; Heart failure; Nonischemic Cardiomyopathy; Multiomics
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples, fasting plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart failure: Adults with heart failure with reduced ejection fraction; no intervention

SUMMARY:
The goal of this observational study is to learn about the composition and function of the gut microbiome in adults with chronic heart failure with reduced ejection fraction. The main questions the study aims to answer are:

1. How does the gut microbiome and its interactions with the host change over time in adults with chronic heart failure?
2. How do these changes relate to heart failure disease severity and complications?

DETAILED DESCRIPTION:
During this study, investigators will recruit adults diagnosed with chronic heart failure with reduced ejection fraction caused by non-ischemic cardiomyopathy. These individuals will undergo longitudinal profiling. This will include detailed profiling of their (1) gut microbiome, (2) blood metabolic and immune markers, and (3) heart failure clinical status. Integrated results will lead to deeper understanding of how gut microbiome interacts with and affects the host in chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction (left ventricular ejection fraction less than 50%)
* Non-ischemic cardiomyopathy
* Body mass index (BMI) 18-40 kg/m2

Exclusion Criteria:

* Treated diabetes
* Advanced kidney disease
* Cirrhosis
* Significant gastrointestinal disease including any history of inflammatory bowel disease
* History of extensive bowel resection
* Active malignancy or systemic chemotherapy within the past 12 months
* Active infection
* Current or recent (within 4 weeks) use of systemic antibiotics, commercial probiotics, immunosuppressive or immunomodulatory medications
* Pregnancy/lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with heart failure with reduced ejection fraction due to non-ischemic cardiomyopathy will be recruited from outpatient cardiomyopathy/heart failure clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Advanced heart failure-associated microbiome signatures | 24 months from baseline visit
  A map of gut microbiome compositional and functional features associated with a composite clinical outcome of advanced heart failure (composite of needing heart transplantation (including active listing), left ventricular assist device implantation, transition to hospice, or death) that occurs within 24 months of baseline visit. Fecal samples will be collected every 3 months over the first 12 month period. Microbiota composition will be determined by shotgun metagenomic sequencing, with taxonomic and metabolic pathway signatures generated using bioinformatic pipelines, respectively. Comprehensive microbiome signatures will encompass alpha and beta diversity, and differential abundance analysis.
Temporal changes in the gut microbiome community composition in chronic heart failure | 12 months from baseline visit
  Longitudinal changes in the gut microbiome composition and functionality in chronic heart failure will be determined. Microbiome signatures will be mapped from fecal samples collected every 3 months over a 12 month period, generated from shotgun metagenomic sequencing data and after processing through bioinformatic pipelines.

SECONDARY OUTCOMES:
Comprehensive longitudinal metabolome profile in chronic heart failure | 12 months from baseline visit
  Changes in the host (human) metabolome profile in chronic heart failure with reduced ejection fraction will be determined. Participants provide fasting blood samples every 3 months for 12 months, from which plasma samples are prepared. Plasma metabolites are run through liquid chromatography-mass spectrometry (LC-MS) columns. MetID (Metabolite Identification from a reference database) and our LC-MS data are used to identify hundreds of metabolites with confidence levels 1-2. Many of the identified metabolites are gut microbiome-derived.
Comprehensive longitudinal cytokine profile in chronic heart failure | 12 months from baseline visit
  Changes in the host (human) cytokines in chronic heart failure with reduced ejection fraction will be determined. Participants provide fasting blood samples every 3 months for 12 months, from which serum samples are prepared. Cytokines are profiled using a 76-cytokine Luminex profiling system at the Stanford Human Immune Monitoring Center. This involves attaching antibodies specific to cytokines to beads using a capture molecule. The fluorescent molecules are attached to the cytokines, and fluorescence is used as the measure of cytokine abundance.
Longitudinal change in New York Heart Association (NYHA) functional class | 12 months from baseline visit
  Participants' functional status (as measured by NYHA class, which ranges from 1 to 4, with 1 being no to minimal symptoms with activity, and 4 being symptoms at rest) will be assessed at each study visit for the first 12 months (every 3 months).
Longitudinal change in the self-reported functional status | 12 months from baseline visit
  Participant self-reported functional status will be assessed via Kansas City Cardiomyopathy Questionnaire-12, which participant will complete at each study visit (every 3 months for 12 months). Overall summary and clinical summary scores (each 0-100, with 0 corresponding to severe and 100 corresponding to no functional limitations) will be calculated and compared over visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data, gut microbiome (taxonomic and metabolic pathway) profiles, plasma metabolome and cytokines (see details below), in addition to analytical code
Supporting Information: Study Protocol, Analytic Code
Time Frame: Immediately upon publication, without end date
Access Criteria: All nucleic acid raw read and processed data will be deposited in Sequence Read Archive (SRA) (metagenomics). Metabolomics and cytokine data will be deposited in Metabolomics Workbench and ImmPort (both of these are National Institutes of Health (NIH) data repositories), respectively. All genomic data sharing will be done in accordance with NIH policies, including the Genomic Data Sharing Policy, and the Institutional Review Board (IRB) approved consent types for each sample type. Detailed metadata will be associated with each dataset. To request access of the data, researchers will use the standard processes at the above repositories. The standard data access processes typically allow access for one year and are renewable. Once the data are submitted to the above repositories, those archive will control the long-term persistence of the data set.